CLINICAL TRIAL: NCT00273208
Title: Being Well, Staying Healthy: An Integrated Mind-Body Medicine Intervention to Decrease Fatigue Among Breast Cancer Survivors, PILOT STUDY
Brief Title: An Intervention to Decrease Fatigue Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MMC 2005-01
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2007-08-02 (Estimated); Status verified 2007-08

CONDITIONS: Fatigue After Adjuvant Breast Cancer Treatment
Keywords: breast cancer; fatigue
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: 10 week behavioral intervention program

SUMMARY:
This research project is being done to design and then test whether a 10 week program can help reduce the symptoms of being tired and fatigued among women who have had breast cancer. The pilot study will include 4 groups of women, two groups of women from Baltimore and two groups of women from Washington County, Maryland. Each group will have 5 to 6 women. The purpose of this pilot study is to help us find the best things to include in the program to help women who have had breast cancer and who have severe problems with fatigue that has lasted months to years after being treated with chemotherapy or radiation therapy.

Following the pilot program we will conduct and evaluate (using a quasi-experimental design comparing fatigue scores before and after the intervention) the efficacy of the refined 10-week integrated mind/body medicine approach to reduce symptoms of fatigue among breast cancer survivors who have completed their adjuvant therapy. Four intervention groups (~12 women per group) will be conducted: two in the urban setting and two in the rural setting. We will assess fatigue symptoms at baseline, immediately after the program, 2 months and 6 months following completion of the program. We will compare mean baseline scores to post-intervention scores.

The ultimate goal is to develop a non-pharmacologic, holistic, low risk intervention for improving symptoms of fatigue and thus improving quality of life among breast cancer survivors

DETAILED DESCRIPTION:
Research Question:

Fatigue is a common, persistent symptom following treatment for breast cancer, challenging a women's ability to promptly regain her overall health and well-being. The aim of the study is to design, evaluate and implement an integrated mind-body medicine intervention to reduce symptoms of persistent fatigue.

The research questions being addressed are: Can a 10 week mind-body medicine intervention program improve fatigue scores from the disability range to the non-disabled range and does the improvement in fatigue symptoms persist up to 6 months following the intervention?

The aims of the study are to Aim I: Pilot test a 10 week mind/body medicine group intervention among 4 groups of breast cancer survivors with 5 women per group. Groups will be stratified by urban/rural setting (Baltimore region/Washington County), race (African American and White), and educational status. These pilot groups will evaluate the program to help refine the intervention to be comprehensible and culturally sensitive.

Aim II: A 10-week intervention program will be developed specifically targeted to alleviate fatigue among breast cancer survivors. Weekly sessions of approximately 2 hours duration will be held. Four intervention groups with approximatley 12 women per group women will be conducted in two regions, an urban setting and a rural setting. The interventions will be conducted at the Women's Center for Health & Medicine at the Mercy Medical Center in downtown Baltimore and the Robinwood Outpatient Medical Facility in Hagerstown Maryland (Washington County.) The Women's center is located downtown Baltimore with access to public transportation as well as a having convenient parking with valet services. The Robinwood Center is also centrally located in Washington County near Hagerstown, MD.

Rationale:

Thirty-five percent of breast cancer survivors, between 1 and 5 years following the diagnosis of breast cancer report symptoms of fatigue that fall into the disability range, despite remaining disease-free (Bower 2000, Lindley 1998). There is a paucity of information on what interventions may be most useful in reducing fatigue symptoms. Most interventions have focused on one factor that may contribute to fatigue such as sleep disturbance or pain. Exercise interventions have been tried but have mostly focused on fatigue during chemotherapy or radiation therapy and have not addressed the problem of persistent fatigue.

Fatigue is a complex, multi-dimensional symptom with several contributing factors. Pain, sleep disturbance, depression, decreased physical activity and menopausal symptoms are associated with fatigue (Couzi 1995, Servaes 2002, Bennett 2004 and Bower 2000). Therefore, a broad-based intervention program holds the most promise for alleviating fatigue. We propose to examine the efficacy of a holistic mind/body medicine approach to empower women to address many of the factors associated with fatigue and incorporate healthy behaviors into their routine to alleviate fatigue. The intervention is a 10 week program modeled after the Mind/Body Medicine program established by Dr. Herbert Benson of the Harvard-affliliated Mind Body Medicine Institute.

Methods Study Design: Quasi-experimental: before/after study design.

Population: The target population is women with breast cancer diagnosed within the past 5 years. The eligibility criteria include:

* Women within 5 years of the diagnosis of breast cancer and currently disease free.
* Women must have completed chemotherapy and/or radiation therapy 6 months prior to joining the study.
* Women may be taking adjuvant hormonal therapy (e.g. tamoxifen or aromatase inhibitors)
* Women scoring less than 50 (consistent with servere fatigue leading to disability and limitations) on the energy/fatigue subscale of the SF-36 health survey (Appendix A).

Intervention:

Each session will last approximately 90 minutes. We will offer the sessions at the most convenient time for participants (e.g. early morning, lunch time or evening). The time will be established based on availability of the participants.

Sample Size:

The pilot study will recruit 5 women for each of 4 groups: Two urban groups, African American and White, and two rural groups, stratified by educational status (less than high school; high school graduate and higher). No formal sample size was calculated for the pilot study. The women will evaluate each session for comprehension and relevance to their situation (e.g. exercise interventions may vary significantly for an urban resident versus a rural resident). Following the completion of the 10 week program we will also ask each woman to evaluate the program as a whole.

Sample size calculations for the main intervention component were based on results of a survey of fatigue and quality of life among breast cancer survivors 1 to 5 years following the diagnosis of breast (Bower 2000). That study used the energy/fatigue subscale of the SF-36 Health Survey (Ware 1992.). That instrument has also been shown to correlate with the Piper fatigue scale, an instrument specifically designed and evaluated among breast cancer patients (Piper 1998). We will administer both survey instruments but will base sample size estimates on the SF-36, a more widely used health survey instrument.

The SF-36 energy/fatigue subscale defines disability/limitation as scores under 50. In a survey of breast cancer survivors, women classified as disabled due to fatigue (scoring less than 50 on the subscale) had a mean score of 37 (Bower 2000.) Overall, in that study, breast cancer survivors had a mean score of 60 (standard deviation 20). Women who fall into the disabled range of the energy/fatigue subscale will be recruited for this study. We estimate that the intervention will improve mean scores to a level of 50/51 (average 14 point improvement) to the non-disabled range. We will compare mean scores before and after the intervention session. Assuming a mean score of 37 and a projected mean score improvement of 14 points 10 women per intervention group will give a power of 80% to detect a mean difference of 14 points (using paired-t-test). We will recruit 12 patients per group, allowing for potential dropouts during the intervention. Thus each of 4 groups of women should provide adequate power to detect a meaningful clinical improvement in fatigue scores.

Recruitment:

Women will be recruited through the Hoffberger Breast Center, the Medical Oncology Practice at Mercy, and, for Washington County, through the John Marsh Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

moderate to severe fatigue >6 months after last chemotherapy or radiation treatment >5 years from diagnosis

-

Exclusion Criteria:

Metastatic disease-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2005-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
change in fatigue score

CONTACTS AND LOCATIONS:
Overall Officials: Kathy J Helzlsouer, M.D., M.H.S., Principal Investigator — Mercy Medical Center
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States